CLINICAL TRIAL: NCT05644795
Title: Efficacy of a Wheat-free Diet in Autoimmune Diseases: a Pilot Therapeutic Study in Sjogren's Disease
Brief Title: Wheat-free Diet in the Treatment of Sjogren's Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: Aurelio Seidita (Unknown)
Responsible Party: Principal Investigator, Pasquale Mansueto, Associate Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACPM31
Record Dates: First submitted 2022-11-09; First posted 2022-12-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sjogren's Syndrome; Non-celiac Gluten Sensitivity
Keywords: Sjogren's Syndrome; Non-celiac Gluten Sensitivity; Non-celiac Wheat Sensitivity
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Population Groups; Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, cross-over, single center clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: wheat/milk free diet (W/MFD) group (Active Comparator): Patients randomized to intervention group will go to a 2 months elimination diet (wheat and cow's milk products). After 2 months of elimination diet they will go to an open challenge, with reintroduction of wheat. After 2 weeks of open diet or whenever rheumatologic, intestinal and/or extraintestinal symptoms should return or intensify, patients will end the study.
  Interventions: Dietary Supplement: Wheat/milk free diet (W/MFD) group
- Placebo Comparator: rice/turkey free diet (R/TFD) group (Placebo Comparator): Patients randomized to control group will go to a 2 months elimination diet (rice and turkey's meat). After 2 months of elimination diet they will crossover to a 2 months elimination diet (wheat and cow's milk products). After 2 months of elimination diet they will go to an open challenge, with reintroduction of wheat. After 2 weeks of open diet or whenever rheumatologic, intestinal and/or extraintestinal symptoms should return or intensify, patients will end the study.
  Interventions: Dietary Supplement: Rice/turkey free diet (R/TFD) group

INTERVENTIONS:
Dietary Supplement: Wheat/milk free diet (W/MFD) group — Patients randomized to intervention diet group will have to follow a wheat and cow's milk products free diet and, after 2 months, they will be exposed to an open wheat challenge, with reintroduction of wheat. After 2 weeks of open diet, or whenever dermatologic, intestinal and/or extraintestinal symptoms should return or intensify, all patients will be revaluated and will end the study.
  Other Names: Intervention Group
  Arms: Active Comparator: wheat/milk free diet (W/MFD) group
Dietary Supplement: Rice/turkey free diet (R/TFD) group — Patients randomized to control diet group will have to follow a diet with elimination of rice and turkey's meat products for 2 months; after that they will crossover to a wheat and cow's milk products free diet and, finally, after 2 months, they will be exposed to an open wheat challenge, with reintroduction of wheat. After 2 weeks of open diet, or whenever dermatologic, intestinal and/or extraintestinal symptoms should return or intensify, all patients will be revaluated and will end the study.
  Other Names: Control Group
  Arms: Placebo Comparator: rice/turkey free diet (R/TFD) group

SUMMARY:
Recent data show that some foods can increase intestinal mucosa permeability and immune activation of subjects with gastrointestinal (GI) symptoms. Wheat seems the most frequent food which activates this inflammatory response and can cause both GI and extra-intestinal symptoms. Patients suffering from wheat-related troubles, in absence of celiac disease diagnosis, can suffer from non-celiac wheat sensitivity (NCWS) and our previous studies showed that about 25% of them are also affected by autoimmune diseases (AD). A gluten-free diet (GFD) can influence inflammatory pattern of AD, including Sjogren's syndrome (SS). Thus, the investigators would enquire if SS patients may also suffer from NCWS and how a wheat-free diet (WFD) modifies their clinical features, and inflammatory and cytokine pattern. The investigators will also assess how wheat reintroduction, by an open challenge, modifies their clinical parameters, intestinal permeability, and both local and systemic inflammatory response.

DETAILED DESCRIPTION:
In recent years, the existence of a wheat-related disorder, in patients who do not suffer from celiac disease (CD) or wheat allergy (WA), has been definitively ascertained and defined as non-celiac wheat sensitivity (NCWS). Its prevalence in the general population is unknown but self-reported NCWS is around 10%. Conflicting data have been reported about the underlying physiopathology. It has been known for years how exposure to gliadin, both in CD and in healthy patients (albeit with reduced levels in the latter), is able to alter intestinal permeability acting on zonulin release and signalling mechanisms. More recently, it has been shown that wheat has high concentrations of wheat amylase-trypsin inhibitors (ATIs), proteins able to activate innate immunity via toll-like receptor-4 (TLR-4) on myeloid cells. Orally ingested ATIs increase intestinal inflammation by activating gut and mesenteric lymphnode myeloid cells.

An increasing number of data have shown that patients with NCWS could have an association with autoimmune diseases, including thyroiditis, undifferentiated connective tissue disease, psoriatic arthritis, spondylarthritis, and Sjogren's syndrome (SS).

SS is an autoimmune disease characterized by an infiltrate of mononuclear cells, mainly lymphocytes, in the exocrine glands, especially the salivary and lacrimal glands. Some preliminary data suggested that a GFD can reduce sialadenitis and increase salivary flow in SS and CD patients. Furthermore, some SS patients have an inflammatory response (release of nitric oxide) to a rectal gluten challenge.

Based on these evidences, as well as on the ability of gluten/wheat to increase intestinal permeability, altering zonulin mechanisms of regulation and signalling, and the ability of some of its components (ATIs, but not only) to activate a local inflammatory response, it could be hypothesized that gluten/wheat may represents one of the pathogenetic environmental factors of SS and that its intake may be able to worsen symptoms in affected patients. In our hypothesis, exposure to gluten/wheat would cause a release of zonulin, which, binding to the surface of the intestinal epithelial cells, is able to modify cell cytoskeleton and to cause the loss of normal occludins function, ultimately leading to an increased monolayer permeability. This increase in permeability would result in greater exposure of the immune system cells to gluten/wheat molecules via activation of TLR-4, with an increase in the infiltration and activation of myeloid cells in the intestinal mucosa and an augmented activity of lymphnode dendritic cells. Such local inflammatory response would have systemic repercussions with alteration of normal cytokine pattern and infiltration of monocytes/macrophages and T cells in the salivary and lacrimal glands, thus being able to contribute, as an environmental factor, to the onset and exacerbation of the clinical manifestations of SS.

Therefore, the investigators hypothesize that a wheat-free diet (WFD) can reduce the inflammatory state and ameliorate the clinical symptoms in SS patients. This hypothesis will be evaluated in both SS patients with associate GI symptoms and in those without GI symptoms. The successive clinical and immunologic reaction to the re-exposure to wheat ingestion, performed by an open challenge, will be also evaluated to confirm a wheat-dependent mechanism and to understand the underlining mechanisms. The project results will provide data about a possible therapeutic role of a WFD in SS and will improve the knowledges about the axis between the intestinal permeability and the systemic inflammation in SS.

More specifically, the investigators aim to:

* identify the prevalence of self-reported NCWS in SS patients;
* assess the overall effect that a WFD plus cow's milk products free diet (CMPFD) determines in symptoms control of the patients affected with SS; the investigators decided to include a CMPFD in association with a WFD because, according to several authors, including our previous studies, NCWS, and more generally gluten-related disorders, are often associated with multiple foods intolerance, first of all cow's milk products intolerance;
* evaluate, by an open wheat challenge, the real frequency of a coexistent NCWS condition;
* assess the possible role played by wheat ingestion in the pathogenesis and molecular mechanisms of SS and NCWS by analysing the variation of intestinal permeability and gut microbiota, in association with cytokines and lymphocytes pattern typical of SS.

ELIGIBILITY:
The study will be a prospective, randomized, placebo-controlled, single center clinical trials. Patients diagnosed with SS, fulfilling the American-European Consensus Group criteria for SS, will be recruited at the outpatient clinic of the Rheumatology Department, University Hospital 'P. Giaccone' of Palermo, Italy.

Inclusion criteria of SS patients

* age >18 and <65 years;
* negativity of anti-deamidated gliadin protein (anti-DGP) immunoglobulins (Ig) class A (IgA) and immunoglobulins (Ig)G, anti-tissue transglutaminase (anti-tTG) class IgA and IgG, and Endomysium antibodies (EmA);
* absence of intestinal villous atrophy, documented in all the patients carrying the DQ2 and/or the DQ8 Human Leukocyte Antigen (HLA) haplotypes (thus irrespective of CD-specific serum antibody negativity
* absence of WA (negative prick-test and/or specific serum immunoglobulin (Ig) E assay for wheat, gluten, and gliadin).

Exclusion criteria of SS patients

* age <18 and >65 years;
* self-exclusion of gluten/wheat from the diet and refusal to reintroduce it, for diagnostic purposes, before entering the study;
* pregnancy;
* alcohol and/or drug abuse;
* Helicobacter pylori and other bacterial and/or parasitic infections;
* diagnosis of chronic inflammatory bowel disease and other organic pathology affecting the digestive system (e.g., severe liver disease), nervous system diseases, major psychiatric disorders, immunological deficits, and impairments that limit physical activity;
* diagnosis of cancer
* patients undergoing chemotherapy and/or radiotherapy.

Study design In a preliminary phase of the study, all patients who access the SS outpatient clinic of the Rheumatology Department of the University Hospital 'P. Giaccone' of Palermo, Italy, will be asked to answer, consecutively, to a questionnaire for the self-assessment of wheat and other foods' intolerance.

After this evaluation, individual's enrollment will start. A database will be predisposed to register demographic, clinical, laboratory, cytofluorimetric and immunohistochemistry data. A repository bank will be used to collect samples from patients at different timepoints.

Patients enrolled based on the inclusion and exclusion criteria and who have agreed to enter the study, after having signed the informed consent, will be randomized, matched for age/gender/racial origin, through a computerized system into an intervention group and a control group. The two groups, each of 15 subjects, will be asked to follow a diet for 2 months. Intervention group will be asked to eliminate wheat and all cow's milk (both fresh and aged) products from the diet (i.e., WFD plus CMPFD). The control group will be asked to eliminate rice and turkey's meat products from the diet. The elimination diet in the control group must be considered as a 'placebo diet' because both rice and turkey's meat are foods known to be used in standard 'oligoantigenic' elimination diet.

Before starting the elimination diet (at time 0, T0), patients will be evaluated by experienced rheumatologists to assess their clinical features, as well as by physicians with expertise in the field of food intolerance about GI and extraintestinal symptoms which could be related to foods intake. Moreover, at this time point, all subjects will be subjected to:

* salivary flux study, by standard sialometry, and salivary samples collection (treated to block enzymatic digestion of proteins), to dose immunologic and inflammatory markers;
* a blood sample, for the analysis of inflammatory markers, cytokine profile, and intestinal permeability markers;
* a urine collection, after the administration of the lactulose/mannitol (LA/MA) test, to define intestinal permeability;
* a collection of stools, for calprotectin assay and definition of the gut microbiota;
* a dietary consult to better explain the dietary approach and provide any information useful to allow adherence to the elimination diet;
* finally, an alimentary (for the self-assessment of adherence to the diet) and symptom's diary will be provided to all patients, which must be filled-in daily.

After 2 months of elimination diet (at time 1, T1), intervention and control patients will be evaluated again both clinically and by laboratory techniques, repeating exactly what have been done at T0. Moreover, they will have to deliver alimentary and symptom's diary, and will discuss the results with physicians.

At this time-point, the subjects enrolled in the intervention group will go to an open challenge, with reintroduction of wheat. After 2 weeks of open diet or whenever rheumatologic, intestinal and/or extraintestinal symptoms should return or intensify (T2int), patients will be valued again both clinically and by laboratory techniques, repeating exactly what have been done at T0 and T1. Patients in this group will end the study at this time-point.

At the same timepoint, patients enrolled in the control group will be asked to repeat the elimination diet, this time removing from the diet wheat and all cow's milk (both fresh and aged) products (i.e., i.e., WFD plus CMPFD, in the context of a cross-over design), for further 2 months (T2con). At the end of these 2 months patients will be valued again both clinically and by laboratory techniques repeating exactly what have been done at T0 and T1. As described before for the intervention group, at this time-point patients of the control group will go to an open challenge with reintroduction of wheat. After 2 weeks of open diet or whenever rheumatologic, intestinal and/or extraintestinal symptoms should return or intensify (T3con), patients will be valued again both clinically and by laboratory techniques repeating exactly what have been done at T0, T1 and T2con. Patients in this group will end the study at this time-point.

Sample size The sample size is difficult to determine as no precise data are known about the effectiveness of a WFD and the response to wheat re-exposure after challenge in SS patients, as well as NCWS frequency in these subjects; previously reported data suggest that about 25% of NCWS patients suffer from an autoimmune disease, and in a study evaluating the effect of a GFD on quality of life, GI symptoms, and immune system in patients with fibromyalgia and NCWS, statistical significance was reached with 10 subjects. Other studies assessing NCWS immunological pattern obtained statistical significance with 26, 30, 22, and 12 patients. Therefore, considering the nature of this prospective and pilot study the investigators planned to enroll a total of 30 patients suffering from SS, 15 with GI symptoms and 15 without, fulfilling the American-European Consensus Group criteria for SS.

Definition of 'positivity' to the open challenge During the open challenge period, patients will be asked to note the possible onset of intestinal and/or extraintestinal symptoms using the food and symptom's diary, using a 10-point Visual Analogic Scale (VAS). The challenges will be stopped when a clinical reaction will occur for at least two consecutive days with a >3-point increase in the patient's recorded symptom VAS scale. The challenges will be considered positive if the same symptoms, which were initially present, will reappear after their disappearance on elimination diet and if the GSRS score and/or the extraintestinal symptoms rating scale will be 25% higher than the same score recorded on elimination diet. Finally, from a strictly rheumatologic point of view, the challenge will be considered positive if a 5% increase in the ESSPRI and ESSDAI score will be registered compared to the same score recorded on the elimination diet.

Statistical Analysis Statistical analysis will be performed using commercial software. Parametric and non-parametric statistical analysis will be performed calculating the mean ± standard deviation (SD) and median, respectively. For comparison of parametric and non-parametric data, the t-test and Mann-Whitney rank-sum test will be used where appropriate. Spearman's correlation analysis will be used to quantify the association between analysed variables. Data will be expressed as mean ± SD. P values less than 0.05 will be considered significant.

All subjects will agree to participate in the study. The study protocol will conform to the ethical guidelines of the Declaration of Helsinki, will be preliminary approved by the Human Research committee of the University Hospital of Palermo, Italy, and registered on the CliniaclTrials.gov. All authors will have access to the study data and will review and approve the final manuscript.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Self-perceived non-celiac wheat sensitivity (NCWS) questionnaire in SS patients | Before enter the study
  To identify SS patients reporting a self-perceived NCWS; all patients will be asked to answer, consecutively, to a validated questionnaire for the self-assessment of wheat and other foods' intolerance. This is a questionnaire self-compiled by patients consisting of three sections: 1) general information (eg. age, sex, highest completed education level, etc.) 2) wheat-related symptoms (sore 0 = no symptoms, score = 1, symptoms after wheat intake; if score = 1 other question qualitatively inquire the symptoms evoked by wheat intake, eg. what kind of symptoms, how long patient perceive this problem, etc.); 3) other foods-related symptoms (score 0 = no symptoms, score 1 = symptoms after intake of other foods; if score = 1 other question qualitatively inquire the symptoms evoked by the intake of the specific food reported by the patients, eg. what kind of symptoms, how long patient perceive this problem, etc.)
Effect of WFD plus CMPFD in symptoms of SS patients as assessed by ESSPRI | From the start of the study (T0) to 2 months of wheat elimination diet (T1).
  To define effects induced by a WFD plus CMPFD in SS patient's symptoms. The following score will be used: European League Against Rheumatism (EULAR) SS Patient Reported Index [ESSPRI, a self-evaluation index measuring symptoms, including pain, fatigue, and dryness, each symptom measured with a single 0, no symptoms, to 10, severe symptoms, scores <5 indicating low and >5 high disease activity).
Effect of WFD plus CMPFD in symptoms of SS patients as assessed by ESSDAI | From the start of the study (T0) to 2 months of wheat elimination diet (T1).
  To define effects induced by a WFD plus CMPFD in SS patient's symptoms. The following score will be used: EULAR SS Disease Activity Index (ESSDAI, a systemic disease activity index, consisting of 12 domains, 11 related to organ involvement and 1 biological domain, cut-off values of >5 and <14 defining moderate, and >14 severe systemic disease activity).
Effect of WFD plus CMPFD in symptoms of SS patients as assessed by GSRS | From the start of the study (T0) to 2 months of wheat elimination diet (T1).
  To define effects induced by a WFD plus CMPFD in SS patient's symptoms. The following score will be used: Gastrointestinal Symptom Rating Scale (GSRS), assessment scale for irritable bowel syndrome-like and functional dyspepsia-like symptoms, providing for a score ranging from 15 (no gastrointestinal symptoms) to 60 (uncontrolled gastrointestinal symptoms).
Effect of WFD plus CMPFD in symptoms of SS patients as assessed by Extraintestinal symptoms rating scale. | From the start of the study (T0) to 2 months of wheat elimination diet (T1).
  To define effects induced by a WFD plus CMPFD in SS patient's symptoms. The following score will be used: Extraintestinal symptoms rating scale, a scoring system based on the symptoms most frequently observed in NCWS patients, providing for a score ranging from 9 (no extra intestinal symptoms) to 34 (uncontrolled extra intestinal symptoms).

SECONDARY OUTCOMES:
Effect of open wheat challenge in symptoms of SS patients as assessed by ESSPRI. | From T1 to 2 weeks of open wheat challenge (T2int and T3con).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in SS patients, both of the intervention group (T2int) and the control group (T3con). The following score will be used: European League Against Rheumatism (EULAR) SS Patient Reported Index [ESSPRI, a self-evaluation index measuring symptoms, including pain, fatigue, and dryness, each symptom measured with a single 0, no symptoms, to 10, severe symptoms, scores <5 indicating low and >5 high disease activity).
Effect of open wheat challenge in symptoms of SS patients as assessed by ESSDAI. | From T1 to 2 weeks of open wheat challenge (T2int and T3con).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in SS patients, both of the intervention group (T2int) and the control group (T3con). The following score will be used: EULAR SS Disease Activity Index (ESSDAI, a systemic disease activity index, consisting of 12 domains, 11 related to organ involvement and 1 biological domain, cut-off values of >5 and <14 defining moderate, and >14 severe systemic disease activity).
Effect of open wheat challenge in symptoms of SS patients as assessed by GSRS. | From T1 to 2 weeks of open wheat challenge (T2int and T3con).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in SS patients, both of the intervention group (T2int) and the control group (T3con). Gastrointestinal Symptom Rating Scale (GSRS), assessment scale for irritable bowel syndrome-like and functional dyspepsia-like symptoms, providing for a score ranging from 15 (no gastrointestinal symptoms) to 60 (uncontrolled gastrointestinal symptoms).
Effect of open wheat challenge in symptoms of SS patients as assessed by Extraintestinal symptoms rating scale. | From T1 to 2 weeks of open wheat challenge (T2int and T3con).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in SS patients, both of the intervention group (T2int) and the control group (T3con). Extraintestinal symptoms rating scale, a scoring system based on the symptoms most frequently observed in NCWS patients, providing for a score ranging from 9 (no extra intestinal symptoms) to 34 (uncontrolled extra intestinal symptoms).
Salivary flux | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Salivary flux (ml/min) will be studied by standard sialometry.
Salivary dosage of immunoglobulin A | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory salivary analysis will be performed to assess immunoglobulin A.
Salivary dosage of immunoglobulin G | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory salivary analysis will be performed to assess immunoglobulin G
Salivary dosage of lactoferrin | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory salivary analysis will be performed to assess lactoferrin.
Salivary dosage of beta 2-microglobulin | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory salivary analysis will be performed to assess beta 2-microglobulin.
Salivary dosage of IL-2 | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory salivary analysis will be performed to assess interleukin (IL)-2
Salivary dosage of IL-6 | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory salivary analysis will be performed to assess interleukin (IL)-6.
Laboratory blood analysis in SS and NCWS patients to assess ESR | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory blood analysis will be performed to assess erythrocyte sedimentation rate (ESR).
Laboratory blood analysis in SS and NCWS patients to assess CRP | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory blood analysis will be performed to assess C-reactive protein (CRP).
Laboratory blood analysis in SS and NCWS patients to assess RF. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory blood analysis will be performed to assess rheumatoid factor (RF).
Laboratory blood analysis in SS and NCWS patients to assess C3 | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory blood analysis will be performed to assess C3
Laboratory blood analysis in SS and NCWS patients to assess C4. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory blood analysis will be performed to assess C4.
Laboratory blood analysis in SS and NCWS patients to assess complete blood count. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory blood analysis will be performed to assess complete blood count.
Laboratory blood analysis in SS and NCWS patients to assess beta 2-microglobulin. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Laboratory blood analysis will be performed to assess beta 2-microglobulin.
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: IL-6
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: IL-10
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: IL-17
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: IL-18
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: IL-21
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: IL-22
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: tumor necrosis factor (TNF)-alpha
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interferon (IFN)-gamma,
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: B cell activating factor (BAF)
Peripheral blood ELISA analysis of inflammatory cytokines in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: C-X-C Motif Chemokine Ligand 13 (CXCL13)
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: lymphocyte T helper (Th)1
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: lymphocyte T helper Th17
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: lymphocyte T helper Th22
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: lymphocyte T regulator (Treg)
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: follicular B helper T cells (Tfh)
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: innate lymphocyte cell (ILC)1
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: innate lymphocyte cell (ILC)2
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: innate lymphocyte cell (ILC)3
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: lymphocyte T cluster of differentiation (CD)8+
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: natural killer (NK) T cells
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern: B cells
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of SS. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of SS pathogenetic pattern:interferon type I signature in cluster of differentiation (CD)14+ monocytes
Peripheral blood ELISA analysis of intestinal permeability markers in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of intestinal permeability markers will be performed to assess: zonulin
Peripheral blood ELISA analysis of intestinal permeability markers in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Peripheral blood ELISA analysis of intestinal permeability markers will be performed to assess: F-Actin
LA/MA test in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Lactulose/Mannitol (LA/MA) test will be performed to assess in vivo intestinal permeability.
Fecal ELISA analysis of inflammatory gut marker in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Fecal ELISA analysis of inflammatory gut marker will be performed to assess fecal calprotectin.
Gut microbiota assessment in SS and NCWS patients. | From the start of the study (T0) to 2 months of wheat elimination diet (T1), to 2 weeks of open wheat challenge (T2int and T3con).
  Gut microbiota assessment will be performed by quantification of gut microbiota on stools samples.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Study Chair — University of Palermo; Giuliana Guggino, MD, Study Chair — University of Palermo
Locations (3):
- Italy (3):
  - Internal Medicine Department of the University Hospital of Palermo, Palermo, Palermo
  - Rheumatology Department of the University Hospital of Palermo, Palermo, PA
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroccio A, Giambalvo O, Blasca F, Iacobucci R, D'Alcamo A, Mansueto P. Self-Reported Non-Celiac Wheat Sensitivity in High School Students: Demographic and Clinical Characteristics. Nutrients. 2017 Jul 19;9(7):771. doi: 10.3390/nu9070771. PMID 28753927
- [Background] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Background] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Background] Fasano S, Mauro D, Macaluso F, Xiao F, Zhao Y, Lu L, Guggino G, Ciccia F. Pathogenesis of primary Sjogren's syndrome beyond B lymphocytes. Clin Exp Rheumatol. 2020 Jul-Aug;38 Suppl 126(4):315-323. Epub 2020 Oct 23. PMID 33095148
- [Background] Rizzo C, Grasso G, Destro Castaniti GM, Ciccia F, Guggino G. Primary Sjogren Syndrome: Focus on Innate Immune Cells and Inflammation. Vaccines (Basel). 2020 Jun 3;8(2):272. doi: 10.3390/vaccines8020272. PMID 32503132
- [Background] Rizzo C, La Barbera L, Lo Pizzo M, Ciccia F, Sireci G, Guggino G. Invariant NKT Cells and Rheumatic Disease: Focus on Primary Sjogren Syndrome. Int J Mol Sci. 2019 Oct 31;20(21):5435. doi: 10.3390/ijms20215435. PMID 31683641